CLINICAL TRIAL: NCT05328453
Title: Prenatal Sonographic 3D VOCAL Thymic Volume Calculation May Predict Intrauterine Growth Restriction
Brief Title: Sonographic 3D Measurement of Fetal Thymus May be Used to Predict the Small Baby in Pregnancy.
Acronym: IUGR
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Guven, Prof. Dr., Karadeniz Technical University
Other Study IDs: 2016/181
Record Dates: First submitted 2022-02-10; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women at 15-24 gestation.: Routine fetal ultrasonography at 15-24 weeks. All sonographic measurements including 3D fetal thymus calculation was measured.
  Interventions: Diagnostic Test: Fetal prenatal ultrasonographic evaluation.

INTERVENTIONS:
Diagnostic Test: Fetal prenatal ultrasonographic evaluation. — Routine fetal ultrasonography at 15-24 weeks. All sonographic measurements including 3D fetal thymus calculation was measured.

SUMMARY:
The exact etiology of intrauterine growth restriction (IUGR) remains unclear but is known to involve immunologic/infectious factors. The thymus is one of the main organs involved in the development of the fetal immune system. The aim of this study was to explore the association between 3D fetal thymus volume (VOCAL) on ultrasound and intrauterine growth restiction by adding the 3-dimensional measurement of thymus volume to the routine fetal ultrasound scan at 15-24 week of gestation.

Investigators performed a prospective clinical study in 100 pregnant women in their second trimester of pregnancy who attended the Fetal Medicine Unit of the Medicine Faculty of Karadeniz Technical University during the study period. Maternal age, gravida, para, BMI, blood pressure, gestational age, BPD, FL ,AC, EFW and fetal timus volume measured with VOCAL programme are recorded. For all patients routine clinical and ultrasound examinations were performed during pregnancy. Gestational age at birth, way of birth and newborn birthweight were recorded. The results were statistically compared in the SPSS 13.0 program. Student-t test and chi-square test were used for statistical analysis. ROC curve analysis was used for limit values. The data of patients with IUGR and without IUGR were compared. The ability of the thymus volume to predict the IUGR was tested using binary logistic regression analysis. P value <0.05 was considered statistically significant.

DETAILED DESCRIPTION:
A signed informed consent form for voluntary participation in the study was provided by all the women. A record was made for each patient of age, gravida, parity, body mass index (BMI), and sonographic measurements of biparietal diameter (BPD), abdominal circumference (AC), femur length (FL), and estimated fetal weight (EFW).

3D Fetal thymus volume (TV) was measured by using a VOLUSON E-10 ultrasonography device, by a single researcher experienced in the use of obstetric ultrasound with a transabdominal volumetric probe. The fetal thymus, transverse section of the fetal chest, and the 3 vessel sections were visualised, then the 3D US modality was activated and the thymus volume was obtained immediately with the same probe.

All cases were followed up in terms of pregnancy complications (IUGR development) until delivery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years,
* Who presented at the polyclinic for routine antenatal follow-up at 15-24 weeks
* Had no complaints.
* Had normal renal, hepatic, and thyroid functions test results.

Exclusion Criteria:

* Any known endocrinopathy,
* systemic disease,
* collagen disorder,
* hypercholesterolemia,
* hemoglobinopathy
* history of neoplasm,
* current or previous cardiovascular disease,
* the use of any drugs within the 3 months before the pregnancy,
* multiple pregnancy,
* current smoking,
* abnormal renal, hepatic, or thyroid function test results,
* the presence of any findings of fetal chromasomal or structural anomaly,
* refusal to participate in the study.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: This prospective cohort study included 100 women with a single pregnancy who presented at the current clinic in one year period and had no risk factors for high-risk pregnancy in the second trimester screening for anomalies.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
IUGR development. | One year period.
  IUGR was accepted as EFW below the 10th percentile according to BPD, FL, and AC

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman Guven, Prof, Study Chair — Karadeniz Technical University Faculty of Medicine Department of Obs and Gyn

IPD SHARING:
Plan to Share IPD: Undecided